CLINICAL TRIAL: NCT01416220
Title: A Randomized, Open-label, Trial of Lithium Versus Paroxetine in Subjects With Major Depression Who Have a Family History of Bipolar Disorder or Completed Suicide
Brief Title: Lithium Versus Paroxetine in Major Depression
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MoodDig-001
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder
Keywords: depression; bipolar disorder; manic depressive illness
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Bipolar Disorder | interventions — Lithium; Lithium Carbonate; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium (Experimental): Following the enrollment period, subjects will enter a six-week randomized treatment period with either lithium or paroxetine. Lithium carbonate will be commenced at 600mgs hs, with increase to 900mgs at day 7. Dose will be flexibly titrated to give a serum level between 0.5 and 1.1mmol/l. At visit 4, the dose of lithium may be adjusted (within the range of 0.6 and 1.1 mmol/l).
  Interventions: Drug: Lithium
- Paroxetine (Active Comparator): Following the enrollment period, subjects will enter a six-week randomized treatment period with either lithium or Paroxetine.Paroxetine will be commenced at 10mgs and increased to 20mgs on day 7.At visit 4, the dose of paroxetine may be increased to 40mgs, if there is no response (less than 20% reduction in MADRS score) as per current Canadian guidelines.
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Lithium — Study drug will be packaged and supplied in an open-label fashion. There will be a washout period of all active psychotropic medication. Psychotropics will be withdrawn over 5 half-lives with the exception of drugs known to cause withdrawal symptoms (primarily antidepressants), which will be tapered over 10 days.
  Following the enrollment period, subjects will enter a six-week randomized treatment period with either lithium or paroxetine. Lithium carbonate will be commenced at 600mgs hs, with increase to 900mgs at day 7. Dose will be flexibly titrated to give a serum level between 0.5 and 1.1mmol/l. At visit 4, the dose of lithium may be adjusted (within the range of 0.6 and 1.1 mmol/l.
  Other Names: lithium carbonate
  Arms: Lithium
Drug: Paroxetine — Study drug will be packaged and supplied in an open-label fashion. There will be a washout period of all active psychotropic medication. Psychotropics will be withdrawn over 5 half-lives with the exception of drugs known to cause withdrawal symptoms (primarily antidepressants), which will be tapered over 10 days.
  Following the enrollment period, subjects will enter a six-week randomized treatment period with either lithium or paroxetine. Paroxetine will be commenced at 10mgs and increased to 20mgs on day 7. At visit 4, the dose of paroxetine may be increased to 40mgs, if there is no response (less than 20% reduction in MADRS score) as per current Canadian guidelines.
  Other Names: paxil
  Arms: Paroxetine

SUMMARY:
This study is being done to look at how well people respond to two different drug treatments for depression. Clinically, people can respond differently to different treatments for reasons which are not always clear. Some research shows that people with a family history of bipolar disorder or completed suicide may react differently to standard medications used to treat depression than those without a family history. The investigators need to know if these drugs are effective to use in patients with depression who have a family history of bipolar disorder or completed suicide.

DETAILED DESCRIPTION:
Lithium is a mood stabilizing drug that has been used to treat people with both bipolar disorder and depression for the last 50 years. It is available to the public by prescription in Canada and has been used by millions of people world wide. Paroxetine is an antidepressant drug that has been used to treat people with depression for the past 10 years. It is also available to the public by prescription in Canada and has been used by millions world wide.

Subjects who join the study, will be given one of the study drugs, either lithium or paroxetine.

Subjects will be randomized "like the flip of a coin" to receive either lithium or paroxetine.

The study drug will be taken once a day by mouth and the daily dose adjusted to find the right dose for the subject. The study drug will be taken for a 6-week period and subjects will be assessed by the research team on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* men or women
* age of 18 years or older
* meet criteria for major depressive episode, and have a family history of bipolar disorder or completed suicide

Exclusion Criteria:

* subjects not able to give informed consent
* pregnant or breast-feeding women
* current panic disorder, post traumatic stress disorder or psychosis
* subjects with a history of mania or hypomania
* subjects with active substance abuse or dependence in the last 6 months
* current depressive episode less than 4 weeks or greater than 12 months in duration
* adequate trial of lithium or paroxetine (lithium level ≥ 0.6mmols/l; paroxetine 20mgs ≥ 5 weeks) for this episode of depression
* concurrent use of other antidepressants or augmenting agents for the treatment of depression
* clinically significant medical illness, in particular renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | Assessed after 6 weeks of treatment
  The primary outcome measure will be reduction in the score on the Montgomery Asberg Depression Rating Scale (MADRS), which has become the standard outcome tool in clinical trials for assessing symptoms of depression. Response will be defined as 50% reduction in MADRS Remission will be defined as MADRS ≤ 12.

SECONDARY OUTCOMES:
The Young Mania Rating Scale (YMRS) | Assessed after 6 weeks of treatment
  This is a standard outcome tool used to assess mania.
The Clinical Global Impression (CGI) | Assessed after 6 weeks of treatment
  The Clinical Global Impression (CGI)is a scale used to measure overall symptom severity, treatment response, and treatment efficacy in patients with mood disorders.
The Columbia Suicide Classification Scale | Assessed over 6 weeks of treatment.
  The Columbia Suicide Classification Scale, used in the FDA analysis of pediatric antidepressants, has become a standard tool used in clinical depression trials and will be used to monitor changes in suicide risk or self-harm weekly.
Barnes Akathisia Rating Scale (BARS) | Assessed over 6 weeks of treatment
  Barnes Akathisia Rating Scale (BARS):
  The BARS is a very brief clinical assessment for the presences of akathisia. Akathisia secondary to antidepressants has been associated with increased suicidality. The inclusion of the BARS will serve to delineate akathisia from psychomotor agitation as part of treatment -emergent mixed symptoms.
Treatment -emergent symptom checklist and questionnaire | Assessed over 6 weeks of treatment
  This checklist and questionnaire will be used to capture a potential range of treatment emergent mixed symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Claire O'Donovan, MD, FRCPC, Principal Investigator — Queen Elizabeth II Health Sciences Centre, CDHA
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada